CLINICAL TRIAL: NCT01162044
Title: Interrupting Traumatic Memories: An Emergency Room Intervention for the Prevention of PTSD
Brief Title: Examining an Emergency Room Intervention for the Prevention of Post Traumatic Stress Disorder (PTSD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr Rena Cooper,, Hadassah Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ER-PTSD-HMO-CTIL
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; prevention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (No Intervention): Subjects will be assessed, but no active intervention given
- Computer game (Experimental): Subjects will play with computer game while in the Emergency Room
  Interventions: Other: Computer game

INTERVENTIONS:
Other: Computer game — Playing with specially designed computer game while in emergency room
  Arms: Computer game

SUMMARY:
PTSD is a common and distressing possible outcome following exposure to a traumatic event. Recent studies show that memory processes may be central to the development of the disorder, and interrupting the consolidation of traumatic memories may prevent the disorder from developing. Specifically the use of a visual spatial task has been shown to reduce a key characteristic of PTSD, intrusions, in non-clinical populations. This study aims to administer a visual spatial task to recent trauma survivors in the Emergency Room, and compare PTSD and symptoms development in these patients as compared to a control group who did not carry out the task. The study hypothesizes that the task will result in less PTSD, lower levels of intrusions, dissociation and pain.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65,
* no loss of consciousness,
* ability to understand study procedures and give informed consent,
* Hebrew as first language,
* experienced a potentially traumatic event as defined in DSM (objective danger and subjective feeling of fear).

Exclusion Criteria:

* current or past psychiatric treatment,
* current or past PTSD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
PTSD symptoms | 6 months
  PTSD status and symptoms as measured by the PSS

CONTACTS AND LOCATIONS:
Overall Officials: Rena Cooper, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel